CLINICAL TRIAL: NCT00780728
Title: Addition of Sildenafil to Bosentan Monotherapy in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Study Evaluating the Addition of Sildenafil to Bosentan Therapy in Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: UHNOHI
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Active Comparator)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil

SUMMARY:
This study will examine the effects of add-on sildenafil to bosentan monotherapy in patients with Pulmonary Arterial Hypertension. Patients on bosentan monotherapy will be followed every 6 months to assess if they have met the pre-defined treatment goals. If a patient fails to achieve these treatment goals or fails to maintain them, sildenafil will be added to their existing bosentan monotherapy. Patients will be assessed 6 months after start of combination therapy for changes in 6MWT, Borg dyspnea scale, WHO functional class, quality of life.

ELIGIBILITY:
Inclusion & Exclusion Criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult